CLINICAL TRIAL: NCT00565916
Title: Role of Estrogen/SERMS on Cardiac Fatty Acid Metabolism (Aim #1- Human Studies)
Brief Title: Evaluating the Roles of Estrogen and Progesterone in Heart Metabolism
Acronym: Estrogen
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Atypically high dropout rate.
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 489; K23HL077179 (NIH); IRB# 04-0812 (Other: IRB); RDRC# 538F (Other: RDRC); GCRC# 966 (Other: GCRC)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Postmenopausal Syndrome
Keywords: Post-Menopausal; PET; Estrogen; Progesterone; Heart Metabolism; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Estrogens; Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- estrogen plus progesterone (Experimental): Hormone replacement therapy (HRT): estrogen plus progesterone
  Interventions: Drug: Estrogen; Drug: Progesterone
- estrogen plus placebo (Active Comparator): Hormone replacement therapy (HRT): estrogen plus placebo
  Interventions: Drug: Estrogen; Drug: Placebo

INTERVENTIONS:
Drug: Estrogen — Estrogen only plus placebo: estradiol topical patch 0.3 mg placed on the lower abdomen for 3 days plus an oral placebo.
  Other procedures: heart metabolism tests which includes a positron-emission tomography (PET) scan, an electrocardiogram (ECG), and an echocardiogram (ECHO).
  Other Names: Estradiol
Drug: Progesterone — Estrogen plus progesterone: estradiol with oral progesterone (Prometrium, 200 mg/day) for 3 days, instead of placebo. Progesterone therapy involves taking a daily oral pill of 200 mg Prometrium for the same 3 days that the estradiol is taken.
  Other Names: prometrium
  Arms: estrogen plus progesterone
Drug: Placebo — Placebo progesterone therapy involves taking a daily placebo pill for the same 3 days that the estradiol is taken.
  Other Names: Inactive Drug
  Arms: estrogen plus placebo

SUMMARY:
Estrogen and progesterone are two main female sex hormones. When a woman goes through menopause, the body's production of estrogen and progesterone significantly decreases. Recent studies have shown that the breakdown of fatty acids in cardiac muscle is important in maintaining a healthy heart, and that estrogen may enhance this process. Also, cardiovascular disease (CVD) occurs more frequently in postmenopausal women than in premenopausal women. This study will determine in postmenopausal women whether estrogen increases the heart's ability to use fats as energy and whether progesterone decreases this effect.

DETAILED DESCRIPTION:
Menopause is a natural event that generally occurs in women between the ages of 45 and 55. During menopause, the body starts producing less estrogen and progesterone until menstruation eventually stops. Estrogen and progesterone are involved in many important functions in a woman's body, and the drastic decline of these hormones in menopause leads to significant changes in the body. Along with such changes, postmenopausal women are at a higher risk than premenopausal women for certain health problems, such as CVD. Previous studies have revealed that alterations in the breakdown of fatty acids in cardiac muscle play a key role in a variety of cardiac disorders. In studies involving human skeletal muscle, estrogen has been shown to increase the breakdown of fatty acids, while progesterone lessens this effect. This study will determine in postmenopausal women whether estrogen increases the heart's ability to break down fats for energy use and whether progesterone decreases this effect. This study will also analyze ovariectomized mice to determine if the candidate specific estrogen receptor modulators (SERMs) raloxifene and tamoxifen increase the heart's ability to use fats as energy and whether the increase is similar to that seen with estrogen. Study investigators will also create estrogen receptor knock-out mice (mice with estrogen receptors removed) to further explore the roles of estrogen and SERMs in heart metabolism.

Participation in this double-blind study will last up to 1 month and will include three study visits. During Visit 1, participants will undergo three standard clinical evaluations. The first evaluation, a medical screening, will include a medical history exam and blood tests to measure estrogen and progesterone levels, liver and kidney function, cholesterol levels, and blood sugar and insulin levels. For the second evaluation, participants will undergo a body composition study to measure total body fat and muscle content using a dual-energy x-ray absorptiometry (DEXA) scan. During the third evaluation, participants will undergo an electrocardiogram (ECG) and an echocardiogram (ECHO), each performed immediately before and after walking on a treadmill. The ECG will measure electrical activity of the heart, and the ECHO will involve imaging the heart with an ultrasound.

Visits 2 and 3, occurring 3 days apart, will each include two imaging tests of the heart: a positron-emission tomographic (PET) scan and a resting ECHO. Throughout both tests an ECG and blood pressure cuff will be used to monitor heart rhythm and blood pressure, respectively. During the PET scan, participants will lie flat in an imaging machine for three 45- to 60- minute intervals. Blood will be drawn and radioactive tracers will be injected via intravenous lines placed in the arms. The ECHO test will also be done during the PET scan.

Between Visits 2 and 3, participants will be randomly assigned to one of two hormone replacement therapy (HRT) regimens: estrogen plus placebo or estrogen plus progesterone. All participants will wear a patch containing estrogen and take a pill of either placebo or progesterone for the 3 days leading up to Visit 3. All participants will be asked for permission to store a sample of their blood for up to 10 years to be used in future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal woman
* Body mass index less than 30
* Practices normal eating habits
* Stops hormone replacement therapy at least 6 months prior to study entry

Exclusion Criteria:

* Currently taking hormone replacement therapy
* History of cardiovascular disease
* Family history of coronary artery disease
* Recent history of smoking, high blood pressure, or hyperlipidemia

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Soto, MD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Castelli WP. Cardiovascular disease in women. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 2):1553-60, 1566-7. doi: 10.1016/0002-9378(88)90189-5. PMID 3377033
- [Background] Bokhari S, Bergmann SR. The effect of estrogen compared to estrogen plus progesterone on the exercise electrocardiogram. J Am Coll Cardiol. 2002 Sep 18;40(6):1092-6. doi: 10.1016/s0735-1097(02)02111-3. PMID 12354433
- [Background] Babiker FA, De Windt LJ, van Eickels M, Grohe C, Meyer R, Doevendans PA. Estrogenic hormone action in the heart: regulatory network and function. Cardiovasc Res. 2002 Feb 15;53(3):709-19. doi: 10.1016/s0008-6363(01)00526-0. PMID 11861041
- [Background] Petrie MC, Dawson NF, Murdoch DR, Davie AP, McMurray JJ. Failure of women's hearts. Circulation. 1999 May 4;99(17):2334-41. doi: 10.1161/01.cir.99.17.2334. No abstract available. PMID 10226101
- [Background] McKee PA, Castelli WP, McNamara PM, Kannel WB. The natural history of congestive heart failure: the Framingham study. N Engl J Med. 1971 Dec 23;285(26):1441-6. doi: 10.1056/NEJM197112232852601. No abstract available. PMID 5122894

RESULTS

PARTICIPANT FLOW:
Groups:
- Hormone Replacement Therapy (HRT): Estrogen Plus Progesterone: Estrogen: HRT with estrogen involves wearing a topical patch of 0.3 mg estradiol. The patch is to be placed on the lower abdomen and worn for 3 days. All participants will also undergo various heart metabolism tests, including a positron-emission tomographic (PET) scan, an electrocardiogram (ECG), and an echocardiogram (ECHO).
  Progesterone: Progesterone therapy involves taking a daily pill of 200 mg Prometrium for the same 3 days that the estradiol is taken.
- Estrogen Plus Placebo: Hormone replacement therapy (HRT): estrogen plus placebo
  Estrogen: HRT with estrogen involves wearing a topical patch of 0.3 mg estradiol. The patch is to be placed on the lower abdomen and worn for 3 days. All participants will also undergo various heart metabolism tests, including a positron-emission tomographic (PET) scan, an electrocardiogram (ECG), and an echocardiogram (ECHO).
  Placebo Progesterone: Placebo progesterone therapy involves taking a daily placebo pill for the same 3 days that the estradiol is taken.
Period: Overall Study
Arm/Group | Hormone Replacement Therapy (HRT): Estrogen Plus Progesterone | Estrogen Plus Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were randomized to receive either estrogen alone, or combined estrogen/projesterone
Groups:
- Estrogen Plus Progesterone: Hormone replacement therapy (HRT): estrogen plus progesterone
  Estrogen: HRT with estrogen involves wearing a topical patch of 0.3 mg estradiol. The patch is to be placed on the lower abdomen and worn for 3 days. All participants will also undergo various heart metabolism tests, including a positron-emission tomographic (PET) scan, an electrocardiogram (ECG), and an echocardiogram (ECHO).
  Progesterone: Progesterone therapy involves taking a daily pill of 200 mg Prometrium for the same 3 days that the estradiol is taken.
- Total: Total of all reporting groups
Arm/Group | Estrogen Plus Progesterone | Estrogen Plus Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had an Increase in Myocardial Fatty Acid Utilization.
Description: Measurements of myocardial fatty acid utilization and oxidation with C[11]-Palmitate and PET in healthy postmenopausal women who take either estrogen alone or with progesterone. The primary outcome measure was designed to determine prospectively whether estrogen will increase the heart's fatty acid utilization and whether progestins will attenuate this effect, in a manner similar to what was seen in an observational study of hormone replacement therapy (HRT) in post-menopausal women. To this end, we had anticipated enrolling 30 healthy post-menopausal women for assessment of cardiac fatty acid metabolism using positron emission tomography (PET) and radioactive C[11]-Palmitate both before and after 3 days of hormone replacement therapy. These volunteers were to be randomized to receive either estrogen alone (E) or combined estrogen/progesterone (EP).
Time Frame: 3 days
Population: 22 healthy post'menopausal women. These volunteers were to be randomized to receive either estrogen alone, or combined estrogen/progesterone. Efforts were made to access the data, PI left institution and there is no access to the data.
Measure: Count of Participants; unit: Participants
Groups:
- Estrogen Plus Progesterone: Hormone replacement therapy (HRT): estrogen plus progesterone
  Estrogen: Estrogen only plus placebo: estradiol topical patch 0.3 mg placed on the lower abdomen for 3 days plus an oral placebo.
  Other procedures: heart metabolism tests which includes a positron-emission tomography (PET) scan, an electrocardiogram (ECG), and an echocardiogram (ECHO).
  Progesterone: Estrogen plus progesterone: estradiol with oral progesterone (Prometrium, 200 mg/day) for 3 days, instead of placebo. Progesterone therapy involves taking a daily oral pill of 200 mg Prometrium for the same 3 days that the estradiol is taken.
- Estrogen Plus Placebo: Hormone replacement therapy (HRT): estrogen plus placebo
  Estrogen: Estrogen only plus placebo: estradiol topical patch 0.3 mg placed on the lower abdomen for 3 days plus an oral placebo.
  Other procedures: heart metabolism tests which includes a positron-emission tomography (PET) scan, an electrocardiogram (ECG), and an echocardiogram (ECHO).
  Placebo: Placebo progesterone therapy involves taking a daily placebo pill for the same 3 days that the estradiol is taken.
Arm/Group | Estrogen Plus Progesterone | Estrogen Plus Placebo
Number analyzed (Participants) | 11 | 11
Participants | NA — PI left institution there is no access to the data. | NA — PI left institution there is no access to the data.

ADVERSE EVENTS:
Time Frame: Per each patient any possible adverse events were collected from the time of consent until the patient completed the study, up to 3 days.
Arm/Group | Estrogen Plus Progesterone | Estrogen Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes